CLINICAL TRIAL: NCT00869856
Title: An Open Label, Single-arm, Baseline-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Immunogenicity of Subcutaneous HX575 Administered Once a Week (qw) and Once Every Two Weeks (q2w) in the Treatment of Anemia Associated With Chronic Kidney Disease in Pre-dialysis and Dialysis Subjects
Brief Title: Study to Evaluate the Efficacy, Safety and Immunogenicity of Subcutaneous HX575 in the Treatment of Anemia Associated With Chronic Kidney Disease (SWEEP)
Acronym: SWEEP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: investigation of adverse events in a related clinical study
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX575-304
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Anemia; Chronic Renal Insufficiency
Keywords: Treatment associated with CRI
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): HX575, EPO Hexal
  Interventions: Drug: HX575 solution for s.c. administration

INTERVENTIONS:
Drug: HX575 solution for s.c. administration — Containing different strengths of epoetin alfa (1 to 10 KIU), s.c. injection, 1x per week (qw) or 1x every two weeks (q2w), injection into abdomen or upper thigh

SUMMARY:
This is an open-label, single-arm, baseline-controlled, multicenter efficacy and safety switch study involving 500 CKD subjects suffering from anemia and treated previously with a stable dose of ESA s.c.

Correction of anemia will be maintained by s.c. administration of HX575 in two frequencies (i.e. qw and q2w), in order to maintain an Hb target range of 10.0-12.0 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Male and female CKD subjects with or without dialysis treatment
* Age > 18 years
* Subjects under documented stable maintenance therapy with ESA, s.c. at least once per week and in accordance with the relevant SmPC, for at least 3 months with a total weekly dose of ≤ 300 IU/kg/week
* Subjects with controlled symptomatic anemia, defined as mean Hb level between 10.0 g/dL and 12.0 g/dL, based on four Hb measurements during the four-week baseline period
* Adequate iron status, serum ferritin ≥ 100 µg/L or transferrin saturation ≥ 20%
* Confirmed negative anti-EPO antibody assay from sample taken at screening visit -4

Exclusion Criteria:

* Systemic cyclosporine
* History of PRCA or aplastic anemia
* History of anti-EPO antibodies
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin level | 36 weeks

SECONDARY OUTCOMES:
To document the safety and lack of immunogenicity of HX575. To determine the optimal dosing regimen of HX575 s.c. administration. | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Roth, Study Chair — Hexal AG
Locations (19):
- Bulgaria (4):
  - MHAT "Dr. Tota Venkova", Gabrovo
  - MHAT Pazardzhik, Pazardzhik
  - MHAT"Sveti Ivan Rilski", Sofia
  - MHAT "Sveta Anna", Varna
- France (2):
  - Polyclinique de Bordeaux-Nord, Bordeaux
  - Centre Hospitalier Universitaire Limoges, Hôpital Dupuytren, Limoges
- Germany (6):
  - KfH Nierenzentrum, Bad König
  - KfH Nierenzentrum, Berlin
  - Gemeinschaftspraxis Dr. Spitthöver, Dr. Knee, Dr. Gröschel, Essen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Gesundheitszentrum Alzey Internistische Gemeinschaftspraxis, Slzrx
  - Nierenzentrum Weinheim Kreiskrankenhaus Weinheim, Weinheim
- Romania (5):
  - Spitalul Clinic de Nefrologie Dr. Carol Davila, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Judetean de Urgenta Deva, Deva
  - Spitalul Clinic Municipal "Dr. Gavril Curteanu", Oradea
  - Spitalul Clinic Judetean Timisoara, Timișoara
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital de Navarra, Pamplona